CLINICAL TRIAL: NCT00008398
Title: A Phase III Study to Test the Efficacy and Safety of GM-CSF to Reduce the Severity and Duration of Mucosal Injury and Pain (Mucositis) Associated With Curative Radiation Therapy in Head and Neck Cancer Patients
Brief Title: Sargramostim in Decreasing Mucositis in Patients Receiving Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: RTOG-9901; CDR0000068406; NCI-P00-0177
Record Dates: First submitted 2001-01-06; First posted 2003-06-05 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Head and Neck Cancer; Oral Complications; Radiation Toxicity
Keywords: stage I nasopharyngeal cancer; stage II nasopharyngeal cancer; stage III nasopharyngeal cancer; stage IV nasopharyngeal cancer; recurrent nasopharyngeal cancer; stage 0 paranasal sinus and nasal cavity cancer; stage 0 nasopharyngeal cancer; stage 0 oropharyngeal cancer; stage 0 laryngeal cancer; stage 0 hypopharyngeal cancer; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; stage 0 lip and oral cavity cancer; stage I lip and oral cavity cancer; stage II lip and oral cavity cancer; stage III lip and oral cavity cancer; stage IV lip and oral cavity cancer; recurrent lip and oral cavity cancer; stage I hypopharyngeal cancer; stage II hypopharyngeal cancer; stage III hypopharyngeal cancer; stage IV hypopharyngeal cancer; recurrent hypopharyngeal cancer; stage I paranasal sinus and nasal cavity cancer; stage II paranasal sinus and nasal cavity cancer; stage III paranasal sinus and nasal cavity cancer; stage IV paranasal sinus and nasal cavity cancer; recurrent paranasal sinus and nasal cavity cancer; stage I oropharyngeal cancer; stage II oropharyngeal cancer; stage III oropharyngeal cancer; stage IV oropharyngeal cancer; recurrent oropharyngeal cancer; oral complications; radiation toxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Hypopharyngeal Neoplasms; Mouth Neoplasms | interventions — sargramostim; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: sargramostim
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Sargramostim may lessen symptoms of mucositis in patients receiving radiation therapy for head and neck cancer. It is not yet known if sargramostim is more effective than no treatment in reducing mucositis caused by radiation therapy.

PURPOSE: Randomized phase III trial to determine the effectiveness of sargramostim in decreasing mucositis in patients who are receiving radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of sargramostim (GM-CSF) in terms of reducing the severity and expected duration of radiotherapy-induced oral mucositis in patients with head and neck cancer receiving radiotherapy.
* Determine the correlation between reduced mucosal injury and quality of life improvement in patients treated with this drug.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to concurrent cisplatin chemotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive radiotherapy once daily five days a week for 6-7 weeks. Patients also receive sargramostim (GM-CSF) subcutaneously (SC) three times a week (except on days if receiving concurrent cisplatin) beginning 1 week prior to radiotherapy and continuing until 2 weeks after completion of radiotherapy for a total of approximately 9 weeks.
* Arm II: Patients receive radiotherapy as in arm I. Patients also receive placebo SC on the same schedule as GM-CSF in arm I.

Quality of life is assessed at baseline, and then at 3, 6, and 12 months.

Patients are followed at 3, 6 and 11 months.

PROJECTED ACCRUAL: A total of 126 patients (63 per arm) will be accrued within 1.2-1.4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed head and neck carcinoma with planned external beam radiotherapy to include 50% of oropharynx, oral cavity, or both]
* Planned external beam radiotherapy of 60-70 Gy total dose to the primary tumor or standard ports for an unknown primary tumor
* Neck metastases from an unknown primary allowed if radiotherapy planned to at least 50% of the salivary gland at a dose of at least 50 Gy
* No T1-T2 glottic tumors
* No residual oral/oropharyngeal injury from prior chemotherapy

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No allergy or idiosyncratic response to sargramostim (GM-CSF)
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No concurrent chemotherapy other than cisplatin

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to the head and neck

Surgery:

* Not specified

Other:

* No concurrent enrollment on other RTOG head and neck studies
* No concurrent oral care medications (e.g., amifostine, chlorhexidrine gluconate, sucralfate, or benzydamine HCl) during study radiotherapy
* No concurrent selective oral cavity decontamination (e.g., IB-367) during study radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-10; Primary Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis G. LeVeque, DDS, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (236):
- United States (217):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscaloosa, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Mount Diablo Medical Center, Concord, California
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Sutter Health West Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center, Pasadena, California
  - Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Inc., San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - St. Joseph's Regional Health System, Stockton, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Saint Mary's Hospital and Medical Center, Grand Junction, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - University of Florida Health Science Center, Gainesville, Florida
  - Edna Williams Cancer Treatment Center, Jacksonville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Clarian Health Partners Inc., Indianapolis, Indiana
  - Regional Cancer Center, Indianapolis, Indiana
  - Oncology Institute of Greater Lafayette, Lafayette, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Lexington Clinic Cancer Center, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - Nebraska Health System, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Radiation Oncology Associates of Albuquerque, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Lourdes Regional Cancer Center, Binghamton, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Finger Lakes Radiation Oncology Center, Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - University of Rochester Cancer Center, Rochester, New York
  - North Shore Radiation Oncology, Setauket, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Regional Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Cancer Center, East Stroudsburg, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Cancer Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon-Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - CCOP - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - All Saints Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (19):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Ryu JK, Swann S, LeVeque F, Scarantino CW, Johnson D, Chen A, Fortin A, Pollock J, Kim H, Ang KK. The impact of concurrent granulocyte macrophage-colony stimulating factor on radiation-induced mucositis in head and neck cancer patients: a double-blind placebo-controlled prospective phase III study by Radiation Therapy Oncology Group 9901. Int J Radiat Oncol Biol Phys. 2007 Mar 1;67(3):643-50. doi: 10.1016/j.ijrobp.2006.09.043. PMID 17293228